CLINICAL TRIAL: NCT07396155
Title: Safety and Efficacy of Allogeneic Umbilical Cord Mesenchymal Stem Cell Therapy in Diabetic Nephropathy Patients: A Clinical Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PT. Prodia Stem Cell Indonesia (Industry)
Collaborators: Dr. Sardjito General Hospital, Yogyakarta, Indonesia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/DN/01/2025
Record Dates: First submitted 2025-07-07; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Nephropathy Type 2
Keywords: Umbilical Cord Mesenchymal Stem Cell; Diabetic Nephropathy; Kidney Disease; Intra-renal Injection; TNF-alpha; IL-10; Glomerular Filtration Rate; eGFR; Regenerative Medicine; Mesenchymal Stem Cells; UC-MSC
MeSH Terms: conditions — Diabetic Nephropathies; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UC-MSC treatment group (Experimental): Participants will receive a single intra-renal injection of UC-MSCs (1 × 10⁶ cells/kg BW), followed by a 12-month monitoring period for safety and renal function outcomes.
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Umbilical Cord Mesenchymal Stem Cells — This intervention consists of a single intra-renal injection of allogeneic umbilical cord-derived mesenchymal stem cells (UC-MSCs) administered under imaging guidance. The dose administered is 1 × 10⁶ cells per kilogram of body weight.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of a single intra-renal injection of allogeneic umbilical cord-derived mesenchymal stem cells (UC-MSCs) in adults with diabetic nephropathy aged 40 to 65 years. The primary questions the study aims to answer are:

1. Is UC-MSC therapy safe and well-tolerated when administered intra-renally in patients with diabetic nephropathy?
2. Does UC-MSC therapy improve kidney function and modulate inflammatory markers over a 12-month follow-up-period?

This is a single-arm, open-label, prospective clinical trial. Participants will receive a one-time intra-renal injection of UC-MSC at a dose of 1 x 10⁶ cells/kg body weight.

Participants will attend scheduled follow-up visits at 1, 3, 6, 9, and 12 months post-injections for evaluation of:

1. Renal function (eGFR, serum creatinine, and urine albumin-creatinine ratio)
2. Inflammatory markers (TNF-α, IL-10)
3. Safety outcomes including early and late adverse events

The results will be compared to baseline measurements to assess changes after the intervention.

If there is a comparison group: Researchers will compare [arm information] to see if [insert effects].

Participants will [describe the main tasks participants will be asked to do, interventions they'll be given and use bullets if it is more than 2 items].

DETAILED DESCRIPTION:
Diabetic nephropathy (DN) is one of the most common microvascular complications of diabetes mellitus and a leading cause of end-stage renal disease worldwide. Despite current standard therapies, many patients continue to experience progressive decline in renal function. As inflammation and immune dysregulation are increasingly recognized as contributors to DN pathogenesis, novel therapeutic strategies targeting these mechanisms are being explored.

Mesenchymal stem cells (MSCs), particularly those derived from umbilical cord tissue, have shown promising anti-inflammatory and regenerative effects in preclinical studies of kidney disease. Their immunomodulatory properties, low immunogenicity, and ease of collection make them a compelling option for cell-based therapies.

This clinical trial aims to evaluate the safety and potential therapeutic benefit of allogeneic umbilical cord-derived MSCs administered via intra-renal injection in individuals with diabetic nephropathy. The study is designed to provide early human data on the feasibility of using UC-MSCs as an adjunctive therapy in DN management. By assessing changes in renal function and inflammatory biomarkers over time, the trial seeks to explore the biological impact of UC-MSC therapy in this population.

This research represents an important step toward developing cell-based interventions for chronic kidney disease, particularly in settings where conventional treatments are insufficient. The findings are expected to contribute valuable data to the growing field of regenerative nephrology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes Mellitus (T2DM)
* Aged between 40 and 65 years
* Diagnosed with chronic kidney disease (CKD) stage III or IV, defined as estimated GFR (eGFR) between 15-60 mL/min/1.73 m² (using CKD-EPI formula)
* Renal biopsy showing diabetic nephropathy type IIa-IV
* Presence of proteinuria, with urine albumin-to-creatinine ratio (UACR) between 30-3000 mg/g (spot morning urine sample)
* Controlled diabetes, defined as HbA1c <10.0% during screening
* Blood pressure within the range of: Systolic 100-160 mmHg, Diastolic 60-100 mmHg
* On stable standard therapy for diabetic nephropathy (e.g. ACE inhibitors or ARBs) for at least 12 weeks prior to screening
* Willing to provide written informed consent and comply with all study procedures until completion

Exclusion Criteria:

* Active malignancy or history of cancer
* Active liver disease or abnormal liver function (ALT or AST ≥2× upper limit of normal)
* Hemoglobin <8 g/dL or platelet count <100,000/µL
* Serious or unstable cerebrovascular or cardiovascular conditions within the last 6 months
* Positive pregnancy test or currently breastfeeding (for women of reproductive age)
* Currently receiving immunosuppressive therapy equivalent to ≥20 mg/day prednisone
* History of participation in other stem cell research or therapy studies

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events and Serious Adverse Events | From baseline up to 12 months post-injection
  Safety is assessed by recording the number and percentage of participants experiencing any adverse events (AEs), including both local and systemic reactions.

SECONDARY OUTCOMES:
Change in Estimated Glomerular Filtration Rate (eGFR) | Baseline and at 1, 3, 6, 9, and 12 months after treatment
  Calculated using the CKD-EPI 2021 formula
Change in Serum Creatinine | Baseline and at 1, 3, 6, 9, and 12 months after treatment
  Measured in mg/dL. Collected via venous blood samples
Change in Urine Albumin-to-Creatinine Ratio (UACR) | Baseline and at 1, 3, 6, 9, and 12 months after treatment
  Measured in mg/g from morning spot urine samples

OTHER OUTCOMES:
Change in Serum TNF-α Levels | Baseline and at 1, 3, 6, 9, and 12 months after treatment
  Tumor necrosis factor-alpha (TNF-α) is measured in patient serum using ELISA as a marker of systemic inflammation. The change in TNF-α concentration from baseline over 12 months will be analyzed to evaluate the immunomodulatory effect of UC-MSC therapy.
Change in Serum IL-10 Levels | Baseline and at 1, 3, 6, 9, and 12 months after treatment
  Interleukin-10 (IL-10) is measured in patient serum using ELISA as an anti-inflammatory cytokine. This outcome assesses whether UC-MSC treatment modulates IL-10 levels over a 12-month follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Sardjito General Hospital, Yogyakarta, Indonesia